CLINICAL TRIAL: NCT04886960
Title: A Phase I/II Randomized Double-Blinded Standard of Care (Corticosteroid) vs. Sterile Amniotic Fluid for Osteoarthritis
Brief Title: pAF for the Treatment of Osteoarthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, David Petron, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 128491
Record Dates: First submitted 2021-04-29; First posted 2021-05-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Osteo Arthritis Knee
Keywords: Amniotic Fluid; Osteo Arthritis
MeSH Terms: interventions — Platelet Activating Factor; MICU1 protein, human; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Half of the patients will be in the SOC treatment arm and half of the patients will be in the AF arm. The PI and patients will be blinded as to the arm in which they will be participating. Once the randomization number is obtained, unblinded research staff will prepare the appropriate study drug. The injections will be blinded to the research coordinator in charge of data entry, the treating physician and the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amniotic Fluid Injection (Experimental): Amniotic Fluid Injection, 3ml, one time dose.
  Interventions: Biological: Amniotic Fluid Injection
- Standard of Care Steroid Injection (Active Comparator): Corticosteroids, 3ml, one time dose.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Biological: Amniotic Fluid Injection — Comparison of Standard of Care (Corticosteroid) injection vs. Sterile Processed Amniotic Fluid Injection for Knee Osteoarthritis
  Other Names: Processed Amniotic Fluid, pAF; Human Amniotic Fluid, hAF
  Arms: Amniotic Fluid Injection
Other: Standard of Care — Comparison of Standard of Care (Corticosteroid) injection vs. Sterile Processed Amniotic Fluid Injection for Knee Osteoarthritis
  Other Names: Corticosteriods 3ml, one time dose
  Arms: Standard of Care Steroid Injection

SUMMARY:
This is a Phase I/II Randomized Double-Blinded Standard of Care (Corticosteroid) vs. Sterile Amniotic Fluid for Osteoarthritis

DETAILED DESCRIPTION:
This study will look at blinded standard of care (SOC) steroid injection vs. amniotic fluid injection (pAF) to treat and reduce osteoarthritis (OA) inflammation and pain. The main objectives of this study are to establish the safety and tolerability of allogeneic intra-articular pAF injections. Secondary objectives include pain levels and functional outcome scoring in patients over a 12 month time frame.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are between the ages of 18-70 years
* A confirmed diagnosis of knee osteoarthritis based on clinical and radiographic findings consistent with Kellgren-Lawrence Stage 2-3 disease
* Patients who have failed conservative treatment (e.g. steroid, activity modification, therapy, etc.) within 3 months
* Unilateral or bilateral chronic knee joint pain >4 months
* Patients who are able to ambulate (i.e. not wheelchair bound)
* Patient reported a typical pain of at least 4 out of 10 during the past week using VAS numeric pain scale (0-10)
* Patients who are of childbearing potential must agree to use adequate contraception for 90 days after study drug injection

Exclusion Criteria:

* Subjects who have had a previous injection (i.e. steroid, platelet rich plasma, or other) within the last 3 months
* A focal chondral defect, defined by x-ray evaluation
* BMI >40 as defined by NIH Clinical Guidelines Body Mass Index
* Concurrent participation in another investigational trial involving systemic administration of agents (within the previous 30 days) or plans to participate in any other allogeneic stem cell therapy trial during the 12 month follow-up period
* Clinical suspicion of infection at injection site
* Any surgeries within 4 weeks, other than diagnostic surgery
* Insulin or self-reported non-insulin dependent diabetic evident of HgA1c ≥8% among known diabetics
* Unable to consent to an English Language Consent Form
* Frank mechanical issues (i.e. locking of the knee)
* Workman's Compensation cases
* Rheumatoid arthritis
* Patients with a known allergy to local anesthetics or components of the study drug (pAF or steroid injection)
* Patients with vascular claudication or neurologic disorders affecting the index lower limb
* Patients with inflammatory arthropathies or connective tissue disorders; or
* Patients with known alcohol or drug abuse or dependence, recreational use of illicit drug or prescription medications, or have used medical marijuana within 7 days of study enrollment
* Patients with history of active cancer/malignancy within 2 years of screening, apart from adequately treated basal cell or squamous cell carcinoma of the skin not associated with the target knee
* Women who are nursing or pregnant
* Patients of childbearing potential who are unwilling to use adequate contraception for 90 days after study drug injection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Repeat allogeneic intra-articular injection within 6 months. | 6 months
  Participants in both the SOC and pAF treatment arms may require and/or request rescue medication (i.e. SOC injection) at any time and will be given per PI discretion as part of standard of care. The clinicians will not know which study arm the study participant is in but will treat the participant with the SOC injection. This information will be documented and collected in the Electronic Medical Record (EMR), as well as the study's electronic data capture system. Participants will not be given any additional pAF injections throughout the study period.
  The participant will continue to be treated with SOC injections as needed. The outcome will be an indicator of whether or not a subject received a rescue medication within 6 months.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 6 months
  Scale 0-100, where higher numbers indicate less problems. The KOOS is a survey that assesses joint symptoms, pain, pain during daily activities, physical function in daily living, as well as physical function during sports or recreational activities.
Visual Analog Scale for pain (VAS Pain) | 6 months
  Scale 0-10, where higher numbers indicate more pain. Pain will be measured by the Visual Analog Scale for pain (VAS Pain). This will consist of a comparison of mean values for VAS scoring scales pre-injection and at the 6 month follow-up assessment. Clinically significant outcomes will be determined based on the minimal clinically important difference (MCID) occurring for each respective scale, which is defined as the smallest reported measurement tool used to quantify perceived level of pain, graded on a scale from 0 to 10 with 0 representing no pain and 10 representing the worse pain possible, and with precise measurement of the marked pain level's distance from 0 comprising the pain level.
Single Assessment Numerical Evaluation (SANE) | 6 months
  Scale 0-100, where higher numbers indicate more pain. The SANE asks the patient to evaluate their percentage of normal on the affected joint of region of interest. This is a one-question survey.
Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function Computer Adaptive Test (PF-CAT) | 6 months
  Scale 0-100, where higher numbers indicate better physical functioning. The PF-CAT is a bank of questions related to physical function. It is a computerized adaptive test that asks the patient to self-report capabilities rather than actual performance of physical activities. It includes functioning of upper extremities, lower extremities, and central regions and also assess instrumental activities of daily living, such as running errands.

OTHER OUTCOMES:
Number of treatment emergent adverse events (AEs) directly related to the injection. | 1 day, 2 days, 1 month, 3 months, 6 months, 12 months
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 1, 3, 6 and 12 months
  Scale 0-100, where higher numbers indicate less problems. The KOOS is a survey that assesses joint symptoms, pain, pain during daily activities, physical function in daily living, as well as physical function during sports or recreational activities.
Visual Analog Scale for pain (VAS Pain). | 1, 3, 6 and 12 months
  Scale 0-10, where higher numbers indicate more pain. Pain will be measured by the Visual Analog Scale for pain (VAS Pain). This will consist of a comparison of mean values for VAS scoring scales pre-injection and at the 6 month follow-up assessment. Clinically significant outcomes will be determined based on the minimal clinically important difference (MCID) occurring for each respective scale, which is defined as the smallest reported measurement tool used to quantify perceived level of pain, graded on a scale from 0 to 10 with 0 representing no pain and 10 representing the worse pain possible, and with precise measurement of the marked pain level's distance from 0 comprising the pain level.
Single Assessment Numerical Evaluation (SANE) | 1, 3, 6 and 12 months
  Scale 0-100, where higher numbers indicate more pain. The SANE asks the patient to evaluate their percentage of normal on the affected joint of region of interest. This is a one-question survey.
Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function Computer Adaptive Test (PF-CAT) | 1, 3, 6 and 12 months
  Scale 0-100, where higher numbers indicate better physical functioning, The PF-CAT is a bank of questions related to physical function. It is a computerized adaptive test that asks the patient to self-report capabilities rather than actual performance of physical activities. It includes functioning of upper extremities, lower extremities, and central regions and also assess instrumental activities of daily living, such as running errands.

CONTACTS AND LOCATIONS:
Overall Officials: David Petron, MD, Principal Investigator — University of Utah Orthopaedic Center
Locations (1):
- University of Utah Orthopedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kotlarz H, Gunnarsson CL, Fang H, Rizzo JA. Insurer and out-of-pocket costs of osteoarthritis in the US: evidence from national survey data. Arthritis Rheum. 2009 Dec;60(12):3546-53. doi: 10.1002/art.24984. PMID 19950287
- [Background] Underwood MA, Gilbert WM, Sherman MP. Amniotic fluid: not just fetal urine anymore. J Perinatol. 2005 May;25(5):341-8. doi: 10.1038/sj.jp.7211290. PMID 15861199
- [Background] Prusa AR, Marton E, Rosner M, Bernaschek G, Hengstschlager M. Oct-4-expressing cells in human amniotic fluid: a new source for stem cell research? Hum Reprod. 2003 Jul;18(7):1489-93. doi: 10.1093/humrep/deg279. PMID 12832377
- [Background] Bottai D, Cigognini D, Nicora E, Moro M, Grimoldi MG, Adami R, Abrignani S, Marconi AM, Di Giulio AM, Gorio A. Third trimester amniotic fluid cells with the capacity to develop neural phenotypes and with heterogeneity among sub-populations. Restor Neurol Neurosci. 2012;30(1):55-68. doi: 10.3233/RNN-2011-0620. PMID 22377907
- [Background] Johnson, H.L., Peritoneal Immunization. The American Journal of Surgery, 1936. 34(2): p. 266-271
- [Background] Shimberg, M., The Use of Amniotic Fluid Concentrate in Orthopedic Conditions. The Journal of Bone and Joint Surgery, 1938(20): p. 167-177
- [Background] Ismail MA, Salti GI, Moawad AH. Effect of amniotic fluid on bacterial recovery and growth: clinical implications. Obstet Gynecol Surv. 1989 Aug;44(8):571-7. doi: 10.1097/00006254-198908000-00001. No abstract available. PMID 2668811
- [Background] Ojo VA, Okpere EE, Obaseiki-Ebor EE. Antimicrobial properties of amniotic fluid from some Nigerian women. Int J Gynaecol Obstet. 1986 Apr;24(2):97-101. doi: 10.1016/0020-7292(86)90002-0. PMID 2874087
- [Background] Siggers J, Ostergaard MV, Siggers RH, Skovgaard K, Molbak L, Thymann T, Schmidt M, Moller HK, Purup S, Fink LN, Frokiaer H, Boye M, Sangild PT, Bering SB. Postnatal amniotic fluid intake reduces gut inflammatory responses and necrotizing enterocolitis in preterm neonates. Am J Physiol Gastrointest Liver Physiol. 2013 May 15;304(10):G864-75. doi: 10.1152/ajpgi.00278.2012. Epub 2013 Mar 21. PMID 23518680
- [Background] Ozgenel GY, Filiz G, Ozcan M. Effects of human amniotic fluid on cartilage regeneration from free perichondrial grafts in rabbits. Br J Plast Surg. 2004 Jul;57(5):423-8. doi: 10.1016/j.bjps.2003.12.021. PMID 15191823
- [Background] Ozgenel GY, Filiz G. Combined application of human amniotic membrane wrapping and hyaluronic acid injection in epineurectomized rat sciatic nerve. J Reconstr Microsurg. 2004 Feb;20(2):153-7. doi: 10.1055/s-2004-820772. PMID 15011124
- [Background] Karacal N, Kosucu P, Cobanglu U, Kutlu N. Effect of human amniotic fluid on bone healing. J Surg Res. 2005 Dec;129(2):283-7. doi: 10.1016/j.jss.2005.03.026. PMID 15916770
- [Background] Castro-Combs J, Noguera G, Cano M, Yew M, Gehlbach PL, Palmer J, Behrens A. Corneal wound healing is modulated by topical application of amniotic fluid in an ex vivo organ culture model. Exp Eye Res. 2008 Jul;87(1):56-63. doi: 10.1016/j.exer.2008.04.010. Epub 2008 Apr 30. PMID 18555991
- [Background] Nyman E, Huss F, Nyman T, Junker J, Kratz G. Hyaluronic acid, an important factor in the wound healing properties of amniotic fluid: in vitro studies of re-epithelialisation in human skin wounds. J Plast Surg Hand Surg. 2013 Apr;47(2):89-92. doi: 10.3109/2000656X.2012.733169. Epub 2013 Jan 29. PMID 23356944
- [Background] Weissenbacher T, Laubender RP, Witkin SS, Gingelmaier A, Schiessl B, Kainer F, Friese K, Jeschke U, Dian D, Karl K. Influence of maternal age, gestational age and fetal gender on expression of immune mediators in amniotic fluid. BMC Res Notes. 2012 Jul 24;5:375. doi: 10.1186/1756-0500-5-375. PMID 22827842
- [Background] Merimee TJ, Grant M, Tyson JE. Insulin-like growth factors in amniotic fluid. J Clin Endocrinol Metab. 1984 Oct;59(4):752-5. doi: 10.1210/jcem-59-4-752. PMID 6384254
- [Background] Hung M, Bounsanga J, Voss MW, Saltzman CL. Establishing minimum clinically important difference values for the Patient-Reported Outcomes Measurement Information System Physical Function, hip disability and osteoarthritis outcome score for joint reconstruction, and knee injury and osteoarthritis outcome score for joint reconstruction in orthopaedics. World J Orthop. 2018 Mar 18;9(3):41-49. doi: 10.5312/wjo.v9.i3.41. eCollection 2018 Mar 18. PMID 29564213
- [Background] Winterstein AP, McGuine TA, Carr KE, Hetzel SJ. Comparison of IKDC and SANE Outcome Measures Following Knee Injury in Active Female Patients. Sports Health. 2013 Nov;5(6):523-9. doi: 10.1177/1941738113499300. PMID 24427427
- [Background] Roos EM, Toksvig-Larsen S. Knee injury and Osteoarthritis Outcome Score (KOOS) - validation and comparison to the WOMAC in total knee replacement. Health Qual Life Outcomes. 2003 May 25;1:17. doi: 10.1186/1477-7525-1-17. PMID 12801417